CLINICAL TRIAL: NCT05753462
Title: Phase 1/2a, Monocentric, Open Label Study to Evaluate the Safety, PK and PD of SQY51 in Paediatric and Adult Patients With a Genetically Confirmed Diagnosis of Duchenne Muscular Dystrophy
Brief Title: Phase 1/2a for Safety, PK and PD of SQY51 in Paediatric and Adult Patients Duchenne Muscular Dystrophy
Acronym: AVANCE1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sqy Therapeutics (Other)
Collaborators: Biotrial (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AVANCE1-1/2a; 2022-500703-49-01 (Other: EMA)
Record Dates: First submitted 2023-02-06; First posted 2023-03-03 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Duchenne; Dystrophin; DMD; Exon skipping; Exon 51; ASO therapeutics; Tricyclo-DNA
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 (Experimental): Participants will receive single escalating doses of 2, 4, 6, 10, 16 and 25 mg/kg by intravenous infusion of SQY51 every 2 weeks.
  Interventions: Drug: Phase 1, SQY51
- Phase 2a - Treatment arm (Dose 1) (Experimental): Non randomized participants will receive by IV dose 1 of SQY51 in 4 blocks of 4-weeks.
  Interventions: Drug: Phase 2a, SQY51 (cohort 1)
- Phase 2a - Treatment arm (Dose 2) (Experimental): Non randomized participants will receive by IV dose 2 of SQY51 in 4 blocks of 4-weeks.
  Interventions: Drug: Phase 2a, SQY51 (cohort 2)
- Phase 2a - Treatment arm (Dose 3) (Experimental): Non randomized participants will receive by IV dose 3 of SQY51 in 4 blocks of 4-weeks.
  Interventions: Drug: Phase 2a, SQY51 (cohort 3)

INTERVENTIONS:
Drug: Phase 1, SQY51 — SQY51 is administered by intravenous infusion.
  Arms: Phase 1
Drug: Phase 2a, SQY51 (cohort 1) — SQY51 is administered by intravenous infusion at dose 1
  Arms: Phase 2a - Treatment arm (Dose 1)
Drug: Phase 2a, SQY51 (cohort 2) — SQY51 is administered by intravenous infusion at dose 2.
  Arms: Phase 2a - Treatment arm (Dose 2)
Drug: Phase 2a, SQY51 (cohort 3) — SQY51 is administered by intravenous infusion at dose 3.
  Arms: Phase 2a - Treatment arm (Dose 3)

SUMMARY:
This is a Phase 1/2a, monocentric, open label study to evaluate the safety, pharmacokinetics, and pharmacodynamics of SQY51 in patients with Duchenne muscular dystrophy

DETAILED DESCRIPTION:
Avance1 is a Phase 1/2a, Monocentric, Open Label Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of SQY51 in 12 patients with a genetically confirmed diagnosis of Duchenne muscular dystrophy, This study will include i) 13-week Phase 1 Multiple Dose Escalation Phase, and a ii) 32-week Phase 2a.

Twelve (12) patients ≥ 6 years, both ambulant and non-ambulant, will be sequentially enrolled in phase 1 and will receive escalating doses of SQY51 once every two weeks. In phase 2a, patients will be allocated in three cohorts in a non-randomized manner.

On the 25th March 2024, SQY Therapeutics received the authorization from the European Medicines Agency (EMA) to initiate the Phase 2a clinical trial. All the patients involved in the Phase 1 will progress to the Phase 2a.

ELIGIBILITY:
INCLUSION CRITERIA FOR PHASE 1:

* Boys of ≥6 years of age and ≥ 16 kg body weight.
* Ambulatory or non-ambulatory status,
* Patients and, if minor, their legal guardians, who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Diagnosed with Duchenne Muscular Dystrophy (DMD), genotypically confirmed with DMD mutations amenable to exon-51 skipping.
* Stable hepatic and renal function.
* Left ventricular ejection fraction (LVEF) at screening ≥40%.
* If clinically indicated, approved concomitant treatment within standards of care guidelines for DMD, such as antihypertensive, vasodilators, lipid lowering, thyroid replacement, vitamins, mineral substitution, gastric protectors, and nutritional supplements.
* Non-invasive mechanical ventilation is permissive if < 16 h/day.
* Being affiliated with a French social security.
* Informed consent form signed by the patient or, if minor, by the legal guardian(s).

INCLUSION CRITERIA FOR PHASE 2a:

Patients must have completed Phase 1 of the study.

EXCLUSION CRITERIA FOR PHASE 1 AND 2a:

* Patient with any serious medical/surgical or psychiatric condition/illness/history that in the opinion of the investigator would jeopardize patient's safety or would interfere with the study assessments/results, including insufficient vaccination against infectious diseases as recommended by national guidelines, medical history of infection with Hepatitis B,C and HIV.
* Patient with any known allergies to products likely to be used in the study (e.g., antiseptics, anesthetics), known hypersensitivity to any of the ingredients, or excipients of the study drug).
* Patient who participated in other investigational study within the last three months, including those with investigational drugs that aim at restoring dystrophin expression such as other antisense oligomers.
* Patient that received gene therapy.
* Patient with intellectual disability or behavioral problem such that they cannot comply with the study procedure.
* Patient with advanced cardiomyopathy and LVEF < 40%. Patients with dysrhythmias and being treated for dysrhythmias. Patients with non-treated tachycardia.
* Patient for which orthopedic surgery is planned during the time of the study.
* Tracheostomized patients and dependent on invasive mechanical ventilation. Non-invasive mechanical ventilation ≥ 16 h/day. Predicted vital forced capacity < 20%. Medical history with more than two respiratory decompensations requiring hospitalization during the previous year. No respiratory decompensation in the four months preceding enrolment.
* Patients on medications that can restore dystrophin expression, tamoxifen and other drugs without indication for DMD or paediatric population.
* Abnormal laboratory values in the clinically significant range.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs in all participants | From baseline up to week 49

SECONDARY OUTCOMES:
Pharmacokinetic plasma concentration of SQY51 (µg/ml) | From baseline up to week 49
Change from baseline in time to rise from floor, time to complete 1-min, 6-min and 10-min walk in ambulant patients as well as MFM and PUL scores in both ambulant and non-ambulant patients | From baseline up to week 49
Changes from baseline in skeletal muscle dystrophin expression | From baseline up to week 49

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Raymond Poincaré, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bladen CL, Rafferty K, Straub V, Monges S, Moresco A, Dawkins H, Roy A, Chamova T, Guergueltcheva V, Korngut L, Campbell C, Dai Y, Barisic N, Kos T, Brabec P, Rahbek J, Lahdetie J, Tuffery-Giraud S, Claustres M, Leturcq F, Ben Yaou R, Walter MC, Schreiber O, Karcagi V, Herczegfalvi A, Viswanathan V, Bayat F, de la Caridad Guerrero Sarmiento I, Ambrosini A, Ceradini F, Kimura E, van den Bergen JC, Rodrigues M, Roxburgh R, Lusakowska A, Oliveira J, Santos R, Neagu E, Butoianu N, Artemieva S, Rasic VM, Posada M, Palau F, Lindvall B, Bloetzer C, Karaduman A, Topaloglu H, Inal S, Oflazer P, Stringer A, Shatillo AV, Martin AS, Peay H, Flanigan KM, Salgado D, von Rekowski B, Lynn S, Heslop E, Gainotti S, Taruscio D, Kirschner J, Verschuuren J, Bushby K, Beroud C, Lochmuller H. The TREAT-NMD Duchenne muscular dystrophy registries: conception, design, and utilization by industry and academia. Hum Mutat. 2013 Nov;34(11):1449-57. doi: 10.1002/humu.22390. Epub 2013 Aug 26. PMID 23913485
- [Background] Ryder S, Leadley RM, Armstrong N, Westwood M, de Kock S, Butt T, Jain M, Kleijnen J. The burden, epidemiology, costs and treatment for Duchenne muscular dystrophy: an evidence review. Orphanet J Rare Dis. 2017 Apr 26;12(1):79. doi: 10.1186/s13023-017-0631-3. PMID 28446219
- [Background] Mendell JR, Shilling C, Leslie ND, Flanigan KM, al-Dahhak R, Gastier-Foster J, Kneile K, Dunn DM, Duval B, Aoyagi A, Hamil C, Mahmoud M, Roush K, Bird L, Rankin C, Lilly H, Street N, Chandrasekar R, Weiss RB. Evidence-based path to newborn screening for Duchenne muscular dystrophy. Ann Neurol. 2012 Mar;71(3):304-13. doi: 10.1002/ana.23528. PMID 22451200
- [Background] Moat SJ, Bradley DM, Salmon R, Clarke A, Hartley L. Newborn bloodspot screening for Duchenne muscular dystrophy: 21 years experience in Wales (UK). Eur J Hum Genet. 2013 Oct;21(10):1049-53. doi: 10.1038/ejhg.2012.301. Epub 2013 Jan 23. PMID 23340516
- [Background] McDonald CM, Henricson EK, Abresch RT, Han JJ, Escolar DM, Florence JM, Duong T, Arrieta A, Clemens PR, Hoffman EP, Cnaan A; Cinrg Investigators. The cooperative international neuromuscular research group Duchenne natural history study--a longitudinal investigation in the era of glucocorticoid therapy: design of protocol and the methods used. Muscle Nerve. 2013 Jul;48(1):32-54. doi: 10.1002/mus.23807. Epub 2013 May 16. PMID 23677550
- [Background] Li D, Mastaglia FL, Fletcher S, Wilton SD. Precision Medicine through Antisense Oligonucleotide-Mediated Exon Skipping. Trends Pharmacol Sci. 2018 Nov;39(11):982-994. doi: 10.1016/j.tips.2018.09.001. Epub 2018 Sep 30. PMID 30282590
- [Background] Echevarria L, Aupy P, Goyenvalle A. Exon-skipping advances for Duchenne muscular dystrophy. Hum Mol Genet. 2018 Aug 1;27(R2):R163-R172. doi: 10.1093/hmg/ddy171. PMID 29771317
- [Background] Goyenvalle A, Griffith G, Babbs A, El Andaloussi S, Ezzat K, Avril A, Dugovic B, Chaussenot R, Ferry A, Voit T, Amthor H, Buhr C, Schurch S, Wood MJ, Davies KE, Vaillend C, Leumann C, Garcia L. Functional correction in mouse models of muscular dystrophy using exon-skipping tricyclo-DNA oligomers. Nat Med. 2015 Mar;21(3):270-5. doi: 10.1038/nm.3765. Epub 2015 Feb 2. PMID 25642938
- [Background] Renneberg D, Leumann CJ. Watson-Crick base-pairing properties of tricyclo-DNA. J Am Chem Soc. 2002 May 29;124(21):5993-6002. doi: 10.1021/ja025569+. PMID 12022832
- [Background] Ittig D, Gerber AB, Leumann CJ. Position-dependent effects on stability in tricyclo-DNA modified oligonucleotide duplexes. Nucleic Acids Res. 2011 Jan;39(1):373-80. doi: 10.1093/nar/gkq733. Epub 2010 Aug 17. PMID 20719742
- [Background] Birnkrant DJ, Bushby K, Bann CM, Apkon SD, Blackwell A, Brumbaugh D, Case LE, Clemens PR, Hadjiyannakis S, Pandya S, Street N, Tomezsko J, Wagner KR, Ward LM, Weber DR; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and neuromuscular, rehabilitation, endocrine, and gastrointestinal and nutritional management. Lancet Neurol. 2018 Mar;17(3):251-267. doi: 10.1016/S1474-4422(18)30024-3. Epub 2018 Feb 3. PMID 29395989
- [Background] Birnkrant DJ, Bushby K, Bann CM, Alman BA, Apkon SD, Blackwell A, Case LE, Cripe L, Hadjiyannakis S, Olson AK, Sheehan DW, Bolen J, Weber DR, Ward LM; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 2: respiratory, cardiac, bone health, and orthopaedic management. Lancet Neurol. 2018 Apr;17(4):347-361. doi: 10.1016/S1474-4422(18)30025-5. Epub 2018 Feb 3. PMID 29395990
- [Background] Birnkrant DJ, Bushby K, Bann CM, Apkon SD, Blackwell A, Colvin MK, Cripe L, Herron AR, Kennedy A, Kinnett K, Naprawa J, Noritz G, Poysky J, Street N, Trout CJ, Weber DR, Ward LM; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 3: primary care, emergency management, psychosocial care, and transitions of care across the lifespan. Lancet Neurol. 2018 May;17(5):445-455. doi: 10.1016/S1474-4422(18)30026-7. Epub 2018 Feb 2. PMID 29398641
- [Background] McDonald CM, Campbell C, Torricelli RE, Finkel RS, Flanigan KM, Goemans N, Heydemann P, Kaminska A, Kirschner J, Muntoni F, Osorio AN, Schara U, Sejersen T, Shieh PB, Sweeney HL, Topaloglu H, Tulinius M, Vilchez JJ, Voit T, Wong B, Elfring G, Kroger H, Luo X, McIntosh J, Ong T, Riebling P, Souza M, Spiegel RJ, Peltz SW, Mercuri E; Clinical Evaluator Training Group; ACT DMD Study Group. Ataluren in patients with nonsense mutation Duchenne muscular dystrophy (ACT DMD): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2017 Sep 23;390(10101):1489-1498. doi: 10.1016/S0140-6736(17)31611-2. Epub 2017 Jul 17. PMID 28728956
- [Background] Mendell JR, Rodino-Klapac LR, Sahenk Z, Roush K, Bird L, Lowes LP, Alfano L, Gomez AM, Lewis S, Kota J, Malik V, Shontz K, Walker CM, Flanigan KM, Corridore M, Kean JR, Allen HD, Shilling C, Melia KR, Sazani P, Saoud JB, Kaye EM; Eteplirsen Study Group. Eteplirsen for the treatment of Duchenne muscular dystrophy. Ann Neurol. 2013 Nov;74(5):637-47. doi: 10.1002/ana.23982. Epub 2013 Sep 10. PMID 23907995
- [Background] Mendell JR, Goemans N, Lowes LP, Alfano LN, Berry K, Shao J, Kaye EM, Mercuri E; Eteplirsen Study Group and Telethon Foundation DMD Italian Network. Longitudinal effect of eteplirsen versus historical control on ambulation in Duchenne muscular dystrophy. Ann Neurol. 2016 Feb;79(2):257-71. doi: 10.1002/ana.24555. Epub 2016 Jan 8. PMID 26573217
- [Background] Charleston JS, Schnell FJ, Dworzak J, Donoghue C, Lewis S, Chen L, Young GD, Milici AJ, Voss J, DeAlwis U, Wentworth B, Rodino-Klapac LR, Sahenk Z, Frank D, Mendell JR. Eteplirsen treatment for Duchenne muscular dystrophy: Exon skipping and dystrophin production. Neurology. 2018 Jun 12;90(24):e2146-e2154. doi: 10.1212/WNL.0000000000005680. Epub 2018 May 11. PMID 29752304
- [Background] Kinane TB, Mayer OH, Duda PW, Lowes LP, Moody SL, Mendell JR. Long-Term Pulmonary Function in Duchenne Muscular Dystrophy: Comparison of Eteplirsen-Treated Patients to Natural History. J Neuromuscul Dis. 2018;5(1):47-58. doi: 10.3233/JND-170272. PMID 29278896
- [Background] Alfano LN, Charleston JS, Connolly AM, Cripe L, Donoghue C, Dracker R, Dworzak J, Eliopoulos H, Frank DE, Lewis S, Lucas K, Lynch J, Milici AJ, Flynt A, Naughton E, Rodino-Klapac LR, Sahenk Z, Schnell FJ, Young GD, Mendell JR, Lowes LP. Long-term treatment with eteplirsen in nonambulatory patients with Duchenne muscular dystrophy. Medicine (Baltimore). 2019 Jun;98(26):e15858. doi: 10.1097/MD.0000000000015858. PMID 31261494
- [Background] Chamberlain JR, Chamberlain JS. Progress toward Gene Therapy for Duchenne Muscular Dystrophy. Mol Ther. 2017 May 3;25(5):1125-1131. doi: 10.1016/j.ymthe.2017.02.019. Epub 2017 Apr 15. PMID 28416280
- [Background] Relizani K, Echevarria L, Zarrouki F, Gastaldi C, Dambrune C, Aupy P, Haeberli A, Komisarski M, Tensorer T, Larcher T, Svinartchouk F, Vaillend C, Garcia L, Goyenvalle A. Palmitic acid conjugation enhances potency of tricyclo-DNA splice switching oligonucleotides. Nucleic Acids Res. 2022 Jan 11;50(1):17-34. doi: 10.1093/nar/gkab1199. PMID 34893881
- [Background] Berard C, Payan C, Hodgkinson I, Fermanian J; MFM Collaborative Study Group. A motor function measure for neuromuscular diseases. Construction and validation study. Neuromuscul Disord. 2005 Jul;15(7):463-70. doi: 10.1016/j.nmd.2005.03.004. PMID 16106528
- [Background] Mayhew AG, Coratti G, Mazzone ES, Klingels K, James M, Pane M, Straub V, Goemans N, Mercuri E; Pul Working Group. Performance of Upper Limb module for Duchenne muscular dystrophy. Dev Med Child Neurol. 2020 May;62(5):633-639. doi: 10.1111/dmcn.14361. Epub 2019 Sep 19. PMID 31538331
- [Background] McDonald CM, Henricson EK, Han JJ, Abresch RT, Nicorici A, Elfring GL, Atkinson L, Reha A, Hirawat S, Miller LL. The 6-minute walk test as a new outcome measure in Duchenne muscular dystrophy. Muscle Nerve. 2010 Apr;41(4):500-10. doi: 10.1002/mus.21544. PMID 19941337
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Servais L, Deconinck N, Moraux A, Benali M, Canal A, Van Parys F, Vereecke W, Wittevrongel S, Mayer M, Desguerre I, Maincent K, Themar-Noel C, Quijano-Roy S, Serari N, Voit T, Hogrel JY. Innovative methods to assess upper limb strength and function in non-ambulant Duchenne patients. Neuromuscul Disord. 2013 Feb;23(2):139-48. doi: 10.1016/j.nmd.2012.10.022. Epub 2012 Dec 5. PMID 23219352
- [Background] Davis SE, Hynan LS, Limbers CA, Andersen CM, Greene MC, Varni JW, Iannaccone ST. The PedsQL in pediatric patients with Duchenne muscular dystrophy: feasibility, reliability, and validity of the Pediatric Quality of Life Inventory Neuromuscular Module and Generic Core Scales. J Clin Neuromuscul Dis. 2010 Mar;11(3):97-109. doi: 10.1097/CND.0b013e3181c5053b. PMID 20215981
- [Background] Rouillon J, Poupiot J, Zocevic A, Amor F, Leger T, Garcia C, Camadro JM, Wong B, Pinilla R, Cosette J, Coenen-Stass AM, Mcclorey G, Roberts TC, Wood MJ, Servais L, Udd B, Voit T, Richard I, Svinartchouk F. Serum proteomic profiling reveals fragments of MYOM3 as potential biomarkers for monitoring the outcome of therapeutic interventions in muscular dystrophies. Hum Mol Genet. 2015 Sep 1;24(17):4916-32. doi: 10.1093/hmg/ddv214. Epub 2015 Jun 9. PMID 26060189
- [Background] McMillan HJ, Gregas M, Darras BT, Kang PB. Serum transaminase levels in boys with Duchenne and Becker muscular dystrophy. Pediatrics. 2011 Jan;127(1):e132-6. doi: 10.1542/peds.2010-0929. Epub 2010 Dec 13. PMID 21149430
- [Background] Spurney CF, Ascheim D, Charnas L, Cripe L, Hor K, King N, Kinnett K, McNally EM, Sauer JM, Sweeney L, Villa C, Markham LW. Current state of cardiac troponin testing in Duchenne muscular dystrophy cardiomyopathy: review and recommendations from the Parent Project Muscular Dystrophy expert panel. Open Heart. 2021 Mar;8(1):e001592. doi: 10.1136/openhrt-2021-001592. PMID 33762424
- [Background] Braat E, Hoste L, De Waele L, Gheysens O, Vermeersch P, Goffin K, Pottel H, Goemans N, Levtchenko E. Renal function in children and adolescents with Duchenne muscular dystrophy. Neuromuscul Disord. 2015 May;25(5):381-7. doi: 10.1016/j.nmd.2015.01.005. Epub 2015 Jan 19. PMID 25683700
- [Background] Filler G, Lepage N. Should the Schwartz formula for estimation of GFR be replaced by cystatin C formula? Pediatr Nephrol. 2003 Oct;18(10):981-5. doi: 10.1007/s00467-003-1271-5. Epub 2003 Aug 13. PMID 12920638